CLINICAL TRIAL: NCT06225375
Title: Prospective Analysis of Flat Polypropylene Mesh in the Treatment of Uterine (by Uterine-sparing Hysteropexy) and Recurrent or Advanced Pelvic Organ Prolapse: a Safety and Feasibility Study
Brief Title: Flat Polypropylene Mesh in the Treatment of Uterine and Recurrent or Advanced Pelvic Organ Prolapse
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan Institution of Women's Health PC (Other)
Responsible Party: Principal Investigator, Salil Khandwala, Medical Director, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20210803
Record Dates: First submitted 2021-08-05; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This will be a single-center, open-label, prospective clinical trial of 30 subjects undergoing pelvic organ prolapse repair using the Restorelle® Flat Mesh in the treatment of uterine (by uterine-sparing hysteropexy) and recurrent or advanced pelvic organ prolapse. They will be followed for a period of 36 months.
  Eligible subjects shall undergo a detailed medical history and physical exam including a Pelvic Organ Prolapse Quantification (POP-Q)13 system assessment to determine the degree of prolapse. Validated self-reported questionnaires will be completed at baseline including the PFDI-20, PFIQ-7, MESA, and PISQ-12. Baseline demographic information shall be documented. A pelvic ultrasound assessment will be performed to assess the pelvic prolapse.
  Subjects shall undergo transvaginal mesh surgery per the surgeon's specifications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment with Restorelle Flat Mesh (Other): Subjects shall undergo transvaginal mesh surgery per the surgeon's specifications. Briefly, a sheet of Restorelle® Flat Mesh-(XL) shall be cut to the dimensions of the former Restorelle® Direct Fix Anterior and Posterior Mesh
  Interventions: Device: Restorelle® Flat Mesh

INTERVENTIONS:
Device: Restorelle® Flat Mesh — Pelvic organ prolapse repair using Restorelle® Flat Mesh

SUMMARY:
This study is being done to evaluate the safety and feasibility of using flat polypropylene Restorelle® mesh, an ultra-lightweight mesh, for transvaginal use in surgically correcting certain specific cases of pelvic organ prolapse, such as recurrent (previous failed native tissue repair), large stage III or IV pelvic organ prolapse, and those with symptomatic uterine prolapse desiring uterine-sparing surgery (called hysteropexy).

DETAILED DESCRIPTION:
This study is being done to evaluate the safety and feasibility of using flat polypropylene Restorelle® mesh, an ultra-lightweight mesh, for transvaginal use in surgically correcting certain specific cases of pelvic organ prolapse, such as recurrent (previous failed native tissue repair), large stage III or IV pelvic organ prolapse, and those with symptomatic uterine prolapse desiring uterine-sparing surgery (called hysteropexy).Subjects shall undergo transvaginal mesh surgery per the surgeon's specifications. The surgical procedure may include either a posterior Restorelle or an anterior Restorelle or a combined anterior and posterior Restorelle based upon the findings of the prolapse.

Briefly, a sheet of Restorelle® Flat Mesh-(XL) shall be cut to the dimensions of the former Restorelle® Direct Fix Anterior and Posterior Mesh The posterior Restorelle® procedure involves a posterior vaginal incision with dissection into the pararectal spaces with attachment of the mesh arms to the sacrospinous ligaments bilaterally. A StatTack™ (Medtronic, Dublin, Ireland) device may be used to affix the mesh to the sacrospinous ligament. The apical portions of the mesh will then be attached to the cervix, with at least two, 2-0 Prolene sutures.

The anterior Restorelle® procedure will be performed through an anterior vaginal incision with dissection into the paravaginal spaces with attachment of the arms to the obturator internus or the proximal arms to the sacrospinous ligaments bilaterally. If the patient has occult stress urinary incontinence on preoperative urodynamic testing, a midurethral sling will be placed. Cystourethroscopy will be systematically performed on all subjects undergoing an anterior repair or a sling procedure. A vaginal oval pessary device may be placed at the end of surgery, and this will stay in for the next few weeks as a vaginal support mold while healing occurs. Surgical details such as operative time, estimated blood loss, and complications will be documented accordingly. Adverse events (both immediate and delayed) will be classified according to severity/seriousness using Clavien-Dindo classification for reporting complications. The timing, resolution, and relatedness of these adverse events to the procedure shall be documented as well.

A clinical examination including vaginal wall retraction will be performed along with a POPQ exam and validated questionnaires at 6 months, 12 months, 24 months, and 36 months from the index surgery. Subjects will also complete a PGI-I assessment which asks, "Compared to how you were doing before your recent pelvic floor surgery, would you say that now you are:" with answers being "much better, a little better, about the same, a little worse, or much worse". Subjects will also complete a survey with questions rating satisfaction/regret with making the decision to proceed with treatment. Additionally a pelvic ultrasound to assess the Restorelle mesh will be performed at these visits. Subjects will also be seen at 1 week , 1 month, 3 months, and 18 months after surgery, and an examination and ultrasound will be performed at these visits, but no study questionnaires will be requested. At each follow-up visit, the subject shall be questioned about de novo pelvic pain, dyspareunia, de novo urinary incontinence, recurrent urinary tract infections, repeat operations or treatments, or other adverse events. A vaginal examination shall be completed to determine any mesh exposures with location, mesh erosions, infection, atypical vaginal discharge, tenderness, retraction or shortening of the vaginal walls, vaginal scarring, fistula formation, de novo vaginal bleeding or granulomas, or hematomas. A bladder scan shall assess for voiding function, and a dipstick urinalysis shall be obtained to determine the presence of cystitis. Based upon subjects' symptoms and results on dipstick urinalysis, urine may also be sent for microscopic urinalysis and culture with sensitivities, and antibiotics may be given.

All CRFs will be kept confidential and maintained by the research coordinator in a locked cabinet. The participants will keep the research team aware of any changes in medical history, and if any adverse effects are detected. Data collected onto a Microsoft Excel spreadsheet. Patient reported measures will be collected on paper forms and data entered into the spreadsheet. Analysis will be conducted after the study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who have completed childbearing,
* Subjects have failed conservative management for POP and desire a surgical option using transvaginal mesh, and who have a:

  1. recurrent vaginal prolapse after a prior failed native tissue repair, OR,
  2. ≥ stage II uterine prolapse where a surgeon would typically perform a hysterectomy if native tissue repair were to be performed, OR,
  3. large pelvic organ prolapse (overall stage of prolapse ≥ stage III) where the risk of recurrence is high if native tissue repair is performed
* Subjects with a uterus desire a uterine-sparing procedure called hysteropexy
* The subject will provide written informed consent acknowledging her desire to participate in the study using transvaginally placed nonabsorbable mesh with the explicit understanding that there are other surgical options available to her, including but not limited to, transabdominal sacrocolpopexy, sacrospinous ligament fixation, and hysterectomy with vaginal wall repair with support.

Exclusion Criteria:

* Subject is unable or unwilling to comply with the follow-up regimen,
* Subject cannot complete study questionnaires,
* Lacks English competency,
* Declines to participate in the investigation,
* Active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI), or tissue necrosis,
* History of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical),
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area,
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months),
* Subject has a systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan syndrome, Ehlers Danlos, collagenosis, polymyositis or polymyalgia rheumatica),
* Chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis,
* Known neurologic or medical condition affecting bladder function (e.g. multiple sclerosis, spinal cord injury, or stroke with residual neurologic deficit),
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis),
* Subject is unable to put her legs up in the dorsal lithotomy position due to hip arthritis,
* Subject is currently participating in or plans to participate in another device or drug study during this study,
* Known sensitivity to polypropylene,
* Previous prolapse repair with mesh in the target compartment(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety outcome | 12 -36 months post operative
  To determine the proportion of subjects with mesh exposures
Primary efficacy outcome | up to 36 months post operative
  To determine the proportion of subjects with surgical success

SECONDARY OUTCOMES:
Adverse events | intraoperative to 36 months
  to determine any intraoperative and postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Salil Khandwala, MD, Principal Investigator — Michigan Women's Institution of health PC.
Locations (1):
- Michigan Women's Institution of Health PC., Dearborn, Michigan, United States